CLINICAL TRIAL: NCT06013085
Title: Effects of Cognitive-behavioral Therapy for Insomnia in Nurses With Post Covid-19 Condition
Acronym: CBT-I
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wen-Chii Tzeng, Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A202205210
Record Dates: First submitted 2023-08-25; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Cognitive Behavioral Therapy
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive behavioral therapy (Experimental): 6 weeks cognitive-behavioral therapy for insomnia
  Interventions: Behavioral: cognitive behavioral therapy
- treat as usual (No Intervention): provide usual care

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — 6 weeks cognitive behavioral therapy
  Arms: cognitive behavioral therapy

SUMMARY:
Background: Neuropsychiatric conditions, such as insomnia, anxiety, depression, and pain are the most common symptoms experienced by nurses after acute infection of COVID-19. Although medication can assist nurses to improve these symptoms simultaneously in a short period of time, they are at risk of overuse of benzodiazepine hypnotics. Previous research supports the usefulness of cognitive behavioral therapy for insomnia (CBT-I) as self-management strategies in adults with insomnia, anxiety, depression, and pain. However, their effects on post COVID-19 condition have not been researched, and no previous head-to-head study compared the effects on these two approaches on insomnia and neuropsychiatric symptoms.

Aim: To investigate the effects of CBT-I on insomnia, anxiety, depression, and pain in nurses with post COVID-19 condition.

Methods: In this two-arm, parallel randomized controlled trial, 100 participants will be 1:1 randomly assigned to one of two groups (CBT-I and control). The intervention phase will last 6 weeks, followed by a three-month follow-up. Primary outcomes are insomnia severity and sleep quality, whereas anxiety, depression, pain, and health-related quality of life are secondary outcomes. These variables will be assessed before and after the intervention, and at 1, 2, and 3 months after the end of the intervention. Additionally, discontinuing benzodiazepine hypnotics will be measured at 3 months after the end of the intervention.

Discussion: This study will provide evidence of the effects of CBT-I on improving insomnia, anxiety, depression, and pain among nurses with post COVID-19 condition. Results could also enhance means by which to discontinue benzodiazepine hypnotics.

ELIGIBILITY:
Inclusion Criteria:

* nurses with post COVID-19 condition

Exclusion Criteria:

* history of sleep apnea, narcolepsy, pregnant, seizure, with pacemaker

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
insomnia severity | 20 weeks
  measured by Insomnia Severity Index before and after the intervention, and at 1, 2, and 3 months after the end of the intervention
sleep quality | 20 weeks
  measured by Pittsburgh Sleep Quality Index
sleep efficiency | 20 weeks
  measured by Fitbit Charge 5

SECONDARY OUTCOMES:
anxiety | 20weeks
  measured by Generalized Anxiety Disorder 7-Item
depression | 20weeks
  measured by Patient Health Questionnaire 9 item
health-related quality of life | 20weeks
  measured by 36-Item Short Form Health Survey

IPD SHARING:
Plan to Share IPD: No
Data available on request due to privacy/ethical restrictions